CLINICAL TRIAL: NCT01040611
Title: Effectiveness of Music Therapy on Anxiety, Depression and Physiological Responses for Inpatients of Tuberculosis
Brief Title: Effectiveness of Music Therapy
Acronym: TMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Chen-Yun Wang, Taipei Municipal Wan Fang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EVA98-13
Record Dates: First submitted 2009-11-17; First posted 2009-12-29 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Tuberculosis
Keywords: music therapy; Tuberculosis; anxiety; physiological response
MeSH Terms: conditions — Tuberculosis; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music therapy (Experimental): This study examined the effectiveness of music therapy on anxiety, depression and physiological responses for patients with tuberculosis.
  Interventions: Behavioral: Music therapy
- Placebo (No Intervention): No music therapy apply to this arm

INTERVENTIONS:
Behavioral: Music therapy — Patients who fit the inclusion criteria were random assigned to either experimental or control group. Patients in experimental group could choose a piece of CD and listen to music with earphone for 30 minutes. Patients in control group just rest for 30 minutes. The procedure was implemented once a day, and sustained for total 5 days.
  Arms: Music therapy

SUMMARY:
Tuberculosis belongs to chronic diseases as a result of the treatment of disease over a long period, admission to negative pressure isolation wards, and restrictions on visitors. During the in-patient admission, patients are vulnerable to social isolation and separation anxiety. If anxiety sustained, patients' quality of life would be affected. Thus, it is important to improve patients' experience of anxiety. Music has the effectiveness of relaxation, and is helpful to patients' anxious status and physiological responses. This study examined the effectiveness of music therapy on anxiety, depression and physiological responses for patients with tuberculosis.

DETAILED DESCRIPTION:
The experimental study was conducted on a medical center of North Taiwan. 66 patients with Tuberculosis were included in this study. Patients who fit the inclusion criteria were randomly assigned to either experimental or control group. Patients in experimental group could choose a piece of CD and listen to music with earphone for 30 minutes. Patients in control group just rest for 30 minutes. The procedure was implemented once a day, and sustained for total 5 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with TB (including patient with drug resistent).
2. Age between 18~65.
3. Conscious Patient without psychiatric/psychological disorders .
4. Patient without Visual, audio disorder.
5. Patient who is able to understand, speak Mandarin and/or Taiwanese, and is able to communicate with written or oral.

Exclusion Criteria:

1. Medical history of psychiatric/psychologic disorder, medication history of anti-anxiety or anti-depressant which might affect mental status.
2. Patient with Visual, audio disorder.
3. Patient who is not comply with 5 day music therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of music therapy on anxiety, depression and physiological responses | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University -WanFang Hospital, Taipei, Taiwan